CLINICAL TRIAL: NCT00525551
Title: Acetylcystein Vid Stapedotomi
Brief Title: Efficacy of Acetylcysteine in Patients Undergoing Surgery for Otosclerosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Karolinska Institutet (Other); AstraZeneca (Industry)
Responsible Party: Principal Investigator, Anders Fridberger, Dr., Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KS-OAS1; EudraCT 2006-006243-31
Record Dates: First submitted 2007-09-04; First posted 2007-09-06 (Estimated); Last update posted 2013-09-11 (Estimated); Status verified 2013-09

CONDITIONS: Otosclerosis
MeSH Terms: conditions — Otosclerosis | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Acetylcysteine
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo (NaCl)

INTERVENTIONS:
Drug: Acetylcysteine — 150 mg / kg body weight. Drug is dissolved in NaCl to a final volume of 300 mL. This volume is infused starting one hour prior to surgery, and continued 1 hour after the end of surgery.
  Arms: 1
Drug: Placebo (NaCl) — 300 mL 0.9% NaCl
  Arms: 2

SUMMARY:
In otosclerosis, one of the tiny bones of the middle ear is unable to move normally. Sounds cannot be transferred to the inner ear and a conductive hearing loss ensues. The disorder is usually treated by an operation where the bone is replaced by a prosthesis. This restores hearing at low sound frequencies. At high frequencies, surgery is less effective. The smaller effect at high frequencies is probably caused by surgically induced inner ear damage.

Animal studies have shown that the drug acetylcysteine can protect the inner ear against damage. It is not known whether the drug has similar effects in humans. This study will assess the efficacy of acetylcysteine in patients undergoing surgery for otosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Otosclerosis where surgery is planned
* Air / bone gap larger than 20 dB
* Normal middle ear status

Exclusion Criteria:

* Hypersensitivity to acetylcysteine
* Deafness on the other ear
* Stapedotomy previously performed on the ear
* Pregnancy
* Asthma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2007-09; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Hearing thresholds | one year

CONTACTS AND LOCATIONS:
Overall Officials: Dan Bagger-Sjoback, M.D.,Ph.D., Study Chair — Karolinska University Hospital; Anders Fridberger, M.D.,Ph.D., Principal Investigator — Karolinska Institutet
Locations (3):
- Sweden (3):
  - Karolinska University Hospital Huddinge, Huddinge
  - Karolinska University Hospital, Dept. of Otorhinolaryngology, Stockholm
  - Academic Hospital, Uppsala

REFERENCES:
- [Derived] Bagger-Sjoback D, Stromback K, Hakizimana P, Plue J, Larsson C, Hultcrantz M, Papatziamos G, Smeds H, Danckwardt-Lilliestrom N, Hellstrom S, Johansson A, Tideholm B, Fridberger A. A randomised, double blind trial of N-Acetylcysteine for hearing protection during stapes surgery. PLoS One. 2015 Mar 12;10(3):e0115657. doi: 10.1371/journal.pone.0115657. eCollection 2015. PMID 25763866